CLINICAL TRIAL: NCT01064765
Title: ACT-HF: Attention, Cognition and Self-Management in Heart Failure
Acronym: ACT-HF
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: Sigma-Tau Research, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 16233A
Record Dates: First submitted 2010-02-03; First posted 2010-02-08 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Heart Failure
Keywords: Heart failure; Self management; cognitive dysfunction; Self management of heart failure
MeSH Terms: conditions — Heart Failure; Cognitive Dysfunction

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart failure: Outpatients with heart failure, age 75 or less, left ventricular ejection fraction 40% or less, english speaking with no known dementia

SUMMARY:
This study is designed to determine if a relationship exists between problems with memory, attention, learning, insight and executive function and self management in heart failure.

DETAILED DESCRIPTION:
Eligible participants are those 75 years of age or less, with left ventricular ejection fractions of 40% or less, english speaking and no known cognitive deficits. Participants will be administered the Repeatable Battery for the Assessment of Neuropsychological Status and the Controlled Oral Word Association test at the study visit. They will also be asked to complete the Self-Care in Heart Failure Index and the Anosognosia Questionnaire for Dementia at their convenience and mail back to investigator. Participants will be contacted in 90 days to determine if they have been hospitalized, and if so, for how many days.

ELIGIBILITY:
Inclusion Criteria:

* 75 years of age or less
* ejection fraction 40% or less
* heart failure 6 months or more
* English speaking
* no known dementia
* no active substance abuse
* presence of caregiver/support

Exclusion Criteria:

* neurologic disorders potentially causing cognitive dysfunction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with history of heart failure 6 months or more meeting inclusion criteria recruited from outpatient clinic who receiving routine care for their heart failure
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2008-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Self-management of heart failure as measured by the Self-Care in Heart Failure Index | at time of enrollment

SECONDARY OUTCOMES:
Duration of hospitalization(s) | 90 days after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Savitri E. Fedson, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States